CLINICAL TRIAL: NCT06346717
Title: The Effect of Mobile Application-Based Care on Functional Status And Self-Care Agency in Patients Undergoing Total Knee Replacement
Brief Title: Mobile Application Based Care for Total Knee Prosthesis Patients
Acronym: KneeMobilApp
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sinop University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SINOPU-elif 2
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Knee Prosthesis; Mobile Application
Keywords: Total Knee Prosthesis; Mobile Application; Nursing Care; Functional Status; Self-Care Power

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): No intervention will be made to the patients in the control group (n = 30). Patients in the control group will receive standard care and discharge education provided by the hospital. Discharge training consists of verbal information about the postoperative period. The "MMD Scale" will be applied to patients who meet the criteria 1 day before the surgery. Patients with a "BCS Scale" ≥ 89 will be included in the study. Patients will be interviewed face to face and written consent will be obtained. Sociodemographic and descriptive data will be obtained with the "Descriptive Patient Form". Discharge day after surgery (3rd day); Functional status level will be measured with KOOS. 3rd and 6th weeks after surgery; Functional status and self-care ability levels will be measured using the KOOS and Self-Care Power Scale, respectively.
- Experimental Group (Experimental): Patients assigned to the intervention group (n=30) will receive "Knee Prosthesis-M" mobile application service for iOS and Android devices, in addition to standard treatment. The "MMD Scale" will first be applied to patients who meet the criteria 1 day before the surgery. Patients with a "BCS Scale" ≥ 89 will be included in the study. Patients will be interviewed face to face and written consent will be obtained. Sociodemographic and descriptive data will be obtained with the "Descriptive Patient Form". The intervention group will also use the "Knee Prosthesis-M" mobile application for 6 weeks, starting from the 1st day of the surgery. Discharge day after surgery (3rd day); The level of functional status will be measured using the KOOS. At the 3rd and 6th weeks after surgery, functional status and self-care skills will be measured using the KOOS and Self-Care Power Scale, respectively.
  Interventions: Behavioral: "Knee Prosthesis-M" mobile application service

INTERVENTIONS:
Behavioral: "Knee Prosthesis-M" mobile application service — In the early phase of mobile application development, qualitative interviews will be conducted with patients with total knee arthroplasty (TKA) experience regarding their own surgery experiences. A training booklet for "Knee prosthesis-M" will be created, taking into account the literature and patient feedback. Then, the "Knee prosthesis-M" application design will be completed. One day before surgery; Written consent will be obtained from patients who meet the criteria via an "Informed Consent Form". Patients in the intervention group will access the "Knee Prosthesis-M" application from their smartphones and will be asked to use it actively for 6 weeks, starting from the 1st day of the surgery. Mobile application-supported care will be provided to the patients by sending information, warning and reminder messages to the patients for 6 weeks.
  Arms: Experimental Group

SUMMARY:
Total knee prosthesis (TKP); It is a surgical treatment used in the management of functional limitations and severe pain occurring on the degenerated joint surface as a result of rheumatoid arthritis, osteoarthritis, posttraumatic arthritis and other nonspecific arthritis. Nursing care is of great importance in the success of TKP surgery. Reducing pain, preventing complications, increasing self-care ability, and improving the quality of life by improving postoperative knee functions are the main goals of postoperative nursing care. In order to achieve these goals, patients and their relatives need to receive training on home care in the post-operative period before discharge. With the increasing use of mobile technologies in daily life and the increasing adoption of e-health, the opportunity for people to improve their self-management skills through e-health is increasing. Mobile Health (m-Health) provides convenience in many areas such as educating the public, warning about potential diseases and disease risks, and communicating with messages, notifications and video when necessary. It also affects the way nursing services are delivered and provides great benefits in the delivery of nursing services. For all these reasons, it was aimed to examine the effect of mobile application-supported care given to patients with total knee prosthesis on functional status and self-care ability.

DETAILED DESCRIPTION:
The population of the research will consist of patients who underwent total knee prosthesis (TKP) surgery in Sinop Atatürk State Hospital Orthopedics and Traumatology Service between March 2024 and March 2025. The sample will consist of a total of 60 patients, 30 patients in the intervention group and 30 patients in the control group, who meet the inclusion criteria for the study. Patients who are 18 years of age or older, literate, have undergone unilateral total knee prosthesis for the first time, have a smartphone, have a score of 89 or above on the "Mobile Learning Readiness (MLD) Scale" and volunteer to participate in the study will be included in the study. Research data will be collected three times: on the day of discharge, 3rd week and 6th week after surgery, using the Descriptive Patient Form, Knee Injury and Osteoarthritis Outcome Score (KOOS) and Self-Care Power Scale. Individuals with TKP in the intervention group will be asked to use the Knee Prosthesis Mobile application (Knee Prosthesis-M) for six weeks. During this process, individuals with TKP in the control group will be ensured to receive standard care. All interviews will be conducted face to face.

ELIGIBILITY:
Inclusion Criteria:

* Who are 18 years or older
* Being literate
* For the first time, unilateral total knee prosthesis was applied
* Having a smart phone
* Scoring 89 or above on the "Mobile learning readiness (MLD) scale"
* Patients who volunteer to participate in the study

Exclusion Criteria:

* Having speech, hearing and visual impairments
* Having a neurological medical diagnosis that affects cognitive status
* Patients with a psychiatric medical diagnosis
* Not using the mobile application at all
* Notification messages are turned off for 72 hours and cannot be reached by phone after this period
* Interrupting communication before data collection processes are completed
* Wanting to leave the study voluntarily

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score = KOOS | one day
  It is a scale used to evaluate symptoms and functional status due to knee injuries and knee osteoarthritis. It has 5 subgroups: pain, other symptoms, functional status in daily living activities, functional status in sports and leisure activities, and knee-related quality of life. It consists of 42 questions that take approximately 10 minutes. A change of 10 points or more on each subscale between 0 and 100 indicates a clinically significant change. It has been reported to have good reliability and validity in patients undergoing joint replacement.

SECONDARY OUTCOMES:
Exercise of Self-Care Agency=ESCA | one day
  The scale is organized as 35 items. The scale is based on four basic features: active and passive response across situations, motivation, knowledge of health practices, and the individual's own feelings and values. Individuals' answers to the self-care power scale were scored from 0 to 4 and evaluated according to the answers given on a 5-point Likert type scale. The answer "It doesn't describe me at all" was given 0 points, the answer "It doesn't describe me much" was given 1 point, the answer "I have no idea" was given 2 points, the answer "It describes me a little" was given 3 points, the answer "It describes me a lot" was given 4 points. There are 8 negative statements (3, 6, 9, 13, 19, 22, 26, 31) in the scale and the scoring is reversed. The highest score obtained from the scale is 140, and an increase in the score indicates that the individual's self-care power increases.

CONTACTS AND LOCATIONS:
Overall Officials: Sonay GÖKTAŞ, PhD, Study Director — Consulting
Locations (1):
- Elif ALTINKAYNAK SARAL, Merkez, Osmaniye Köyü, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No